CLINICAL TRIAL: NCT06634290
Title: Influence of Cemented Cephalic Augmentation on the Outcome of Osteosynthesis Using Intramedullary Nailing in the Surgical Treatment of Pertrochanteric Hip Fractures in the Elderly
Brief Title: Influence of Cemented Cephalic Augmentation on the Outcome of Intramedullary Nailing in Pertrochanteric Hip Fractures
Acronym: HipOsGal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diego Matías Domínguez Prado (Other)
Responsible Party: Sponsor-Investigator, Diego Matías Domínguez Prado, Specialist in Orthopedic Surgery and Traumatology, PhD, Fundacin Biomedica Galicia Sur
Organization: Fundacin Biomedica Galicia Sur (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-235
Record Dates: First submitted 2024-09-11; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hip Fracture of Intertrochanteric Type
Keywords: hip fracture; osteosynthesis; intramedullary nailing; bone cement augmentation
MeSH Terms: conditions — Hip Fractures | interventions — Fracture Fixation, Internal; Fracture Fixation, Intramedullary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cemented (Experimental): Patients diagnosed of pertrochanteric hip fracture treated with intramedullary nailing WITH cephalic augmentation using bone cement
  Interventions: Device: intramedullary nailing augmentation
- Not Cemented (Active Comparator): Patients diagnosed of pertrochanteric hip fracture treated with intramedullary nailing WITHOUT cephalic augmentation
  Interventions: Device: intramedullary nailing

INTERVENTIONS:
Device: intramedullary nailing augmentation — Treatment of pertrochanteric hip fractures with intramedullary nailing with cephalic augmentation with bone cement
  Other Names: Osteosynthesis
  Arms: Cemented
Device: intramedullary nailing — Treatment of pertrochanteric hip fractures with intramedullary nailing without cephalic augmentation
  Other Names: osteosynthesis
  Arms: Not Cemented

SUMMARY:
The goal of this clinical trial is to learn if small modifications in the surgical technique for the treatment of some kind of hip fractures, improve the result of the surgery. This small modification includes the addition of surgical bone cement to part of the intramedullary nail used in the surgery, to find out if it provides more stability to the construct and represents an improvement in the surgery result.

The main question it aims to answer is:

Does the addition of bone cement produces a decrease in complications related to mechanical failure of the implant used in the surgery and a decrease in the need for re-operation?

Researchers will compare adding this bone cement to the standard surgical technique without it.

Patients will:

* Be randomly assigned to a group that will have surgery following standard protocol or to a group that will have surgery following standard protocol but adding bone cement to the construct.
* Receive standard care for these fractures during hospitalization and posterior follow-up checkups for a year.

DETAILED DESCRIPTION:
Hypothesis

The hypothesis of the study assumes that cephalic augmentation with polymethylmethacrylate cement of the intramedullary nail in the surgical treatment of pertrochanteric hip fractures due to fragility, produces a decrease in complications in relation to mechanical failure of the implant and a decrease in the re-operation rate.

Objectives

The main objective seeks to compare the mechanical failure rates of the implant between intramedullary nailing with and without cephalic augmentation with polymethylmethacrylate cement.

The secondary objectives are to compare the perioperative, 1-month, and 1-year mortality rates of patients treated with intramedullary nailing with and without cephalic augmentation and to evaluate the safety of the surgical technique.

Design

For these purposes, a multicenter, controlled, randomized, single-blind, parallel groups, clinical trial will be carried out.

Participants

Patients over 75 years old, diagnosed with pertrochanteric hip fracture due and requiring surgical intervention, will be eligible for inclusion in the study. All patients will receive surgical treatment using the intramedullary nailing technique, which is the current gold standard treatment for this type of fractures.

Recruitment

Almost all patients who suffer a hip fracture require urgent attention for this process, as well as hospital admission. From the first moment of admission through the emergency room or during the time of hospitalization prior to surgery, the patient and/or their legal representative, will receive pertinent information about the diagnosis, prognosis and treatment of this pathology by and Orthopedic Surgeon.

At the same time that they receive this information, either the principal investigator, or one of the collaborating researchers, will additionally provide information about the study and will recruit patients to participate in it. Prior to the surgery, informed consent will be granted to participate in the research study and the corresponding documents will be signed, along with the usual surgical informed consent used in each institution for this specific pathology,

Given the characteristics of this pathology and the benefit it represents in terms of functional recovery and improved survival, if the surgical intervention is performed in the first 48 hours from the occurrence of the fracture, in some of the patients participating in the study, it may be the case that the operation is performed in less than 24 hours from the acceptance and signing of the informed consent.

Randomization

The patients included in the study will be randomly distributed into two groups, experimental and control. The experimental or CEMENT group will include patients treated with intramedullary nailing WITH cephalic augmentation, and the control or NO CEMENT group will include patients treated with intramedullary nailing WITHOUT cephalic augmentation. Once participation in the study has been accepted and the informed consents have been signed, the randomization process will proceed in the different groups as follows.

The use of a centralized computer system that generates the randomization sequence and performs the registration of the participants, concealment of the randomization sequence and group allocation, is currently the most recommended procedure for conducting clinical trials. For this study, the OxMaR computer system (acronym for Oxford Minimization and Randomization) was used. Each investigator will assign a code to each recruited patient that is recorded in the online randomization form, along with the type of fracture and the patient's sex, which are included as minimization variables.

Description of the intervention

Once the participants have been recruited for the study and have been randomly assigned to the experimental or control group, the surgical intervention will be carried out following the principles of usual clinical practice.

The patient will be operated by an orthopedic surgeon hospital following the usual protocol of the hospital and surgical technique. The implant used will be in all cases an intramedullary nail. Depending on whether the patient has been included in the experimental or control group, surgery will be performed by adding augmentation with polymethylmethacrylate cement to the cephalic component or not.

Regarding blinding, the patient will remain blind to the assignment to one group or another and only the surgeon and the researchers will know the group to which they have been assigned to, given that cement augmentation is easily identifiable for them in a standard radiological control taken during follow-up.

The rest of the follow-up will follow the usual clinical practice during hospital admission and subsequently on an outpatient basis, with controls in outpatient clinics at one month, three months, six months and one year post-intervention. A radiological control will be taken in all follow-ups. Both the clinical follow-up by the surgeon and the radiological follow-up are the same as those carried out in normal clinical practice for this type of pathology. No greater number of visits, consultations, complementary tests, procedures or additional participation are required from the patient for participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* 75 years of age or older.
* Diagnosis with a pertrochanteric fragility fracture.
* Informed consent for participation in the study.

Exclusion Criteria:

* Not meeting the inclusion criteria described above.
* Refusal of the patient or his/her legal representative to participate in the study.
* Diagnosis with hip fracture of subtypes other than 31A1, 31A2, 31A3 and 31B3 of AO-OTA classification.
* Bilateral hip fractures in the same episode.
* Suffering from previous medical pathologies or comorbidities that contraindicate surgical intervention and indicate conservative management of the fracture.
* Performing a surgical technique different from intramedullary nailing or using a surgical implant different from that used in the present study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Mechanical failure rate of the implant | From date of surgery until the date of mechanical failure diagnosis, assessed up to 52 weeks
  Defined as the intolerable loss of reduction of the fracture and the failure of osteosynthesis due to breakage or disassembly of the implant used, which requires surgical reintervention.

SECONDARY OUTCOMES:
Perioperative mortality rate | From date of surgery until the date of hospital discharge, assessed up to a maximum of 7 days
  Proportion of participants who die compared to the total participants during hospital stay, assessed up to a maximum of 7 days
One-month mortality rate | From date of surgery up to 30 days
  Proportion of participants who die compared to the total participants during a period of 30 days
One-year mortality rate | From date of surgery up to 52 weeks
  Proportion of participants who die compared to the total participants during a period of 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diego Matias Dominguez Prado, MD, PhD, Principal Investigator — Complexo Hospitalario de Ourense
Locations (6):
- Spain (6):
  - Hospital de Monforte de Lemos, Monforte de Lemos, Lugo
  - Hospital de Verin, Verín, Ourense
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital do Salnes, Vilagarcía de Arousa, Pontevedra
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Complexo Hospitalario Pontevedra, Pontevedra

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD. Anonymized.
Supporting Information: Study Protocol, ICF
Time Frame: Starting 3 months after publication of results
Access Criteria: Researchers who wish to access data for meta-analysis. Data sharing must be approved by principal research who can be contacted by e-mail.